CLINICAL TRIAL: NCT00180973
Title: MULTICENTRIC INTERNATIONAL RANDOMIZED PHASE III TRIAL COMPARING, NEOADJUVANT CHEMOTHERAPY FOLLOWED BY STANDARD RADIOTHERAPY VERSUS THE SAME NEOADJUVANT CHEMOTHERAPY FOLLOWED BY STANDARD RADIOTHERAPY ASSOCIATED WITH DAILY HYDROXYUREA IN THE TREATMENT OF LOCALLY ADVANCED UNDIFFERENTIATED CARCINOMA NASOPHARYNGEAL TYPE.
Brief Title: PHASE III TRIAL COMPARING, NEOADJUVANT CHEMOTHERAPY FOLLOWED BY STANDARD RADIOTHERAPY VERSUS THE SAME NEOADJUVANT CHEMOTHERAPY FOLLOWED BY STANDARD RADIOTHERAPY ASSOCIATED WITH DAILY HYDROXYUREA IN THE TREATMENT OF LOCALLY ADVANCED UNDIFFERENTIATED CARCINOMA NASOPHARYNGEAL TYPE.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VUMCA2; CSET 94/346
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: LOCALLY ADVANCED UNDIFFERENTIATED CARCINOMA NASOPHARYNGEAL TYPE UCNT
MeSH Terms: interventions — Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea

SUMMARY:
MULTICENTRIC INTERNATIONAL RANDOMIZED PHASE III TRIAL COMPARING, NEOADJUVANT CHEMOTHERAPY (BEC REGIMEN) FOLLOWED BY STANDARD RADIOTHERAPY (70 Gy / 7 WEEKS) VERSUS THE SAME NEOADJUVANT CHEMOTHERAPY FOLLOWED BY STANDARD RADIOTHERAPY ASSOCIATED WITH DAILY HYDROXYUREA IN THE TREATMENT OF LOCALLY ADVANCED UNDIFFERENTIATED CARCINOMA NASOPHARYNGEAL TYPE (UCNT).

ELIGIBILITY:
Inclusion Criteria:

* of either sex
* aged *15 and * 70 years
* never previously treated with radiotherapy, chemotherapy or surgery for malignant disease (except neck adenectomy/diagnosis)
* with aWHO performance status * 2.
* amenable to regular follow-up
* capable of receiving chemotherapy and radiotherapy : in particular, with no contraindications to the use of anthracyclines, bleomycin or cisplatinum.
* with informed consent at entry time, in writing or witnessed oral informed consent, in accordance with local legislation requirements.
* Laboratory requirement : *Baseline hematologic status :

Neutrophil count * 2000 /mm3 Platelet count * 150,000 /mm3 Hemoglobin * 10 g / dl

Exclusion Criteria:

* Histologic types other than type II - III of the WHO classification
* T1 - T2 N0 - N1 or patients with metastatic
* Aged < 15 or > 70.
* Patients in whom chemotherapy is contraindicated: history of myocardial infarction over the last 6 months before inclusion, or clinically present cardiac pathology.
* WHO Performance status >2
* History of prior malignancies (other than non melanoma skin cancer or excised cervical carcinoma in situ).
* Uncontrolled infection,
* Patients refusing participation.
* Patients who, for social, familial or geographic reasons are unlikely to comply with a long term follow-up.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 520
Dates: Start 1995-02

PRIMARY OUTCOMES:
5 year overall survival rate

SECONDARY OUTCOMES:
Time to progresion and local control at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: François ESCHWEGE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France